CLINICAL TRIAL: NCT06726447
Title: sAItisfACES - Impact of an Artificial Intelligence Tool on the Satisfaction of Professionals and Patients in Ambulatory Consultations: A Randomized Cluster Study
Brief Title: Artificial Intelligence Satisfaction in Professionals and Patients
Acronym: sAItisfACES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Dr. in Pain Research, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: sAItisfACES - IA satisfaction
Record Dates: First submitted 2024-11-26; First posted 2024-12-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: General Health Status
Keywords: Artificial Intelligence; Patient Satisfaction; Medical Records Systems, Computerized; Health Care Quality, Access, and Evaluation
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Clusters
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The masking is single-blind and patient-centered, which is appropriate for this type of intervention where it is not feasible to blind healthcare professionals. This helps to reduce bias in measurements related to patient satisfaction and experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence Tool (Experimental): The health centers assigned to this group will implement an artificial intelligence (AI) tool for clinical registration during outpatient consultations. Healthcare professionals will activate the tool at the beginning of the consultation and deactivate it at the end. The tool will be used to document interactions in real time, generating more detailed records and reducing the administrative burden.
  Interventions: Device: Artificial Intelligence Tool
- Standard of care (No Intervention): In the centers assigned to this group, consultations will be carried out in the usual way, using traditional clinical recording methods, without additional technological intervention. This group will serve as a reference to compare differences in satisfaction, duration of consultations and quality of the clinical record.

INTERVENTIONS:
Device: Artificial Intelligence Tool — The intervention in this study consists of the implementation of an artificial intelligence tool for clinical registration during outpatient consultations. This technology facilitates the documentation of interactions in real time, optimizing the workflow of professionals and enabling more patient-centered care.
  Arms: Artificial Intelligence Tool

SUMMARY:
This multicenter cluster-randomized study evaluates the impact of an artificial intelligence (AI) tool on the satisfaction of healthcare professionals and patients in outpatient consultations, measuring its effect on perceived satisfaction (through a visual analog scale), the duration of consultations, and the quality and quantity of clinical data recorded. Adult patients (18-80 years) seen in outpatient centers will participate, comparing those using the AI tool with centers following the usual procedure. The tool is expected to reduce the administrative burden, improve user satisfaction and increase the efficiency and quality of the clinical registry. Recruitment will take place between December 2024 and May 2025, with final analysis planned for the end of 2025.

DETAILED DESCRIPTION:
This multicenter cluster-randomized study aims to evaluate the impact of an artificial intelligence (AI) tool designed to optimize real-time clinical registration during outpatient consultations. Its effect on patient and healthcare professional satisfaction will be analyzed, measured using a visual analog scale (VAS) and validated tools such as the Patient Experience Questionnaire (PEQ) and the Net Promoter Score (NPS). In addition, the duration of consultations and the quantity and quality of clinical data recorded in the intervention and control groups will be compared. The intervention group will use the AI tool, while the control group will continue with the usual recording without AI. Participants will be adult patients (18-80 years) seen in health centers linked to the study, recruited by prior informed consent. AI is expected to reduce the administrative burden on professionals, allowing them to devote more time to direct care, improving both the quality of the clinical record and the patient experience. Recruitment will take place between December 2024 and May 2025, and will follow the ethical guidelines set out in the Declaration of Helsinki. This project seeks to provide evidence on the implementation of AI-based technologies in the outpatient setting and their impact on the quality of healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years of age.
* Patients consulting for any health reason in the outpatient clinics of the centers participating in the study.
* Patients who sign the informed consent to participate in the study.

Exclusion Criteria:

* Patients who are unable to understand or complete the questionnaires, due to:
* Language barriers.
* Cognitive disabilities.
* Any other reason that prevents their adequate participation.
* Patients who are currently participating in other clinical trials or research studies that may interfere with the results of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the consultation | From enrrolment to the end of the consultation the same day.
  measured using a 10 cm Visual Analog Scale (VAS) of satisfaction, which assesses the degree of satisfaction perceived by patients and health professionals. From no satisfaction in the left side to Completely satisfied in the right side.

SECONDARY OUTCOMES:
Duration of the consultation | From enrrolment to the end of the consultation the same day.
  Total time of the consultation, measured manually from the time of entry to the time of departure of the patient.
Number of clinical data recorded | From enrrolment to the end of the consultation the same day.
  Total number of words documented in the clinical history generated during the consultation, excluding headings
Patient Experience (Patient Expectation Questionnaire - PEQ) | at the begining and at the end of the consultation
  Assessment of selected domains of the Patient Expectation Questionnaire (Health Service Process and Professional-Patient Communication). Format: 5-point Likert scale.
Likelihood of recommendation (Net Promoter Score - NPS) | From enrrolment to the end of the consultation the same day.
  Patient's assessment of the likelihood of recommending the service received. Range: 0 (very unlikely) to 10 (very likely).

OTHER OUTCOMES:
Sociodemographic variables | at the begining of the consultation, Just after enrrollment.
  Age (years)
Sociodemographic variables | at the begining of the consultation, Just after enrrollment.
  Sex (Male/Female)
Sociodemographic variables | at the begining of the consultation, Just after enrrollment.
  Nationality (Spanish/Other).
Sociodemographic variables | at the begining of the consultation, Just after enrrollment.
  Municipality of residence (Rural/Non-rural).
Sociodemographic variables | at the begining of the consultation, Just after enrrollment.
  Marital status (Single, Married, Divorced, Widowed).
Sociodemographic variables | at the begining of the consultation, Just after enrrollment.
  Employment status (Active/Not active/Pensioner/Employed/Other).
Sociodemographic variables | at the begining of the consultation, Just after enrrollment.
  Educational level (None, Primary, Secondary, Vocational training, University, Doctorate).

CONTACTS AND LOCATIONS:
Overall Officials: Raul Ferrer, PhD, Principal Investigator — Senior Lecturer and Investigator
Locations (2):
- Spain (2):
  - ACES Centers, Barcelona, Catalonia
  - CSEU La Salle - UAM, Madrid

IPD SHARING:
Plan to Share IPD: No
The study data will not be shared to ensure the confidentiality and privacy of the participants, in accordance with current regulations such as the General Data Protection Regulation (GDPR). In addition, sensitive health-related data are handled, the disclosure of which could compromise the privacy of individuals. Although the data will be anonymized, the team has decided to limit its access to authorized personnel only in order to protect the integrity of the study and minimize ethical or legal risks associated with the distribution of personal information.

REFERENCES:
- [Background] Topol EJ. High-performance medicine: the convergence of human and artificial intelligence. Nat Med. 2019 Jan;25(1):44-56. doi: 10.1038/s41591-018-0300-7. Epub 2019 Jan 7. PMID 30617339